CLINICAL TRIAL: NCT03429400
Title: A Multicenter, Open-Label, Safety and Pharmacokinetic Study of Oral Morphine Sulfate Administration in Pediatric Subjects 2 Years Old Through 17 Years Old With Postoperative Pain
Brief Title: Study of Oral Morphine Sulfate Administration in Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West-Ward Pharmaceutical (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORP-OS+T-(2-17)-SPK-2
Record Dates: First submitted 2018-01-18; First posted 2018-02-12 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Morphine Sulfate (Other): oral morphine sulfate tablets oral morphine sulfate oral solution
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — Morphine every 4 hours as needed for up to a maximum of 5 days

SUMMARY:
This is a multicenter, open-label study to evaluate the safety and PK of oral morphine sulfate in pediatric subjects with post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Has a parent or guardian providing written parental permission/informed consent, with subject assent (if required by local IRB).
2. Has an age-appropriate pain score of ≥4 prior to receiving first dose of study drug.
3. Is a child 2 years old through 17 years old, inclusive (at the time of informed consent signing).
4. Weighs at least 10 kg.
5. Has a routine pediatric procedure that is expected to require inpatient hospitalization postoperatively.
6. Must be an inpatient for the study treatment period.
7. Is expected by the investigator to have moderate to severe postoperative pain requiring the use of oral opioids for treatment.
8. Has the ability to read and understand the study procedures and has the ability to communicate meaningfully with the study investigator and staff (if the subject is of preverbal age or cannot read or communicate meaningfully, then the subject's parent or guardian must meet this criterion).
9. Is able to tolerate oral medications within 48 hours of surgery.
10. If female subject is of childbearing potential, she must have a negative urine pregnancy test result on the day of surgery prior to surgery. In this population, female of childbearing potential is defined by the onset of menarche, ie, menstruation, whether at irregular or regular intervals (periods).
11. Female subjects of childbearing potential and male subjects with partners capable of reproduction must agree to use an effective contraceptive method as follows from the time of Screening through 30 days after the last dose of study drug:

    * A highly effective method of contraception, including hormonal contraceptives (eg, combined oral contraceptives, patch, vaginal ring, injectables, and implants), intrauterine device or intrauterine system OR
    * An effective double-barrier contraceptive method (2 of the following: male condom, female condom, cervical cap, diaphragm, or contraceptive sponge) OR
    * Abstinence
12. Must have vascular access to facilitate blood draws.

Exclusion Criteria:

1. Has significant medical disease(s), laboratory abnormalities, or conditions(s) that in the investigator's judgment could compromise the subject's welfare, ability to communicate with study staff, complete study activities, or would otherwise contraindicate study participation. There is no minimum value for SpO2 for inclusion in the study; this should be based on the investigator's judgment.
2. Has used opioids chronically (eg, codeine, morphine, oxycodone, or hydromorphone), for >7 calendar days within the previous 30 days prior to surgery.
3. Has received codeine, hydrocodone, morphine or oxycodone in any form in the previous 7 calendar days prior to surgery.
4. Is undergoing procedure for treatment of acute burns.
5. Has known hypersensitivity or contraindication to receiving oral opioid(s).
6. Has a current active enteral malabsorption disorder.
7. Has impaired liver function (eg, alanine aminotransferase [ALT] ≥3 times the upper limit of normal [ULN], or total bilirubin ≥2 times ULN [except patients with evidence of Gilbert's syndrome]), known active hepatic disease (eg, hepatitis), evidence of clinically significant chronic liver disease or other condition affecting the liver (eg, chronic hepatitis) that may suggest the potential for an increased susceptibility to hepatic toxicity with oral morphine exposure. Subjects with no previous history of liver function impairment may be enrolled prior to receipt of screening laboratory testing results.
8. Has significantly impaired renal function or disease, as evidenced by an estimated glomerular filtration rate (ie, from creatinine levels using the Schwartz formula) calculated to be less than one-third of normal for the applicable age of this study population. Subjects with no previous history of kidney function impairment may be enrolled prior to receipt of screening laboratory testing results.
9. Has a history of substance abuse or there is evidence of current substance abuse, in the investigator's opinion.
10. Has received epidural or regional anesthesia within 12 hours prior to the first dose of study drug.
11. Has participated in an interventional clinical study (investigational or marketed product) within 30 days before screening, or plans to participate in another clinical trial in the next 30 days.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Measurement of Maximum Plasma Concentration [Cmax] | 24 hours
  Eight PK samples will be collected within the first 24 hours after the first dose
Measurement of Area Under the Curve [AUC] | 24 hours
  Eight PK samples will be collected within the first 24 hours after the first dose
Number of Subjects who experience any AEs that lead to study discontinuation | 6 days
Number of subjects who experience serious adverse events | 6 days
Number of subjects with a UMSS sedation score of 4 | 6 days

SECONDARY OUTCOMES:
Number of subjects who experience any AEs of special interest | 6 days
  AEs of special interest include but not limited to sedation, respiratory depression, nausea, vomiting, and pruritus of moderate-to-severe intensity/grade
Percentage of subjects with clinically significant decreases in SpO2 | 6 days
Number of subject who experience significant change in respiratory rate | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Schmidt, MD,PhD, Study Director — Premier Research
Locations (1):
- Site 105, Sheffield, Alabama, United States